CLINICAL TRIAL: NCT04474015
Title: Optimizing Volunteer Comfort for Transcranial Electrical Stimulation (TES): An Assessment of Sensor (Electrode) Preparations - PARTS A, B and C
Brief Title: Optimizing Volunteer Comfort for Transcranial Electrical Stimulation (TES): An Assessment
Acronym: TES
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: WRAIR #1927
Record Dates: First submitted 2019-11-12; First posted 2020-07-16 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Performance Enhancing Product Use; Sleep

STUDY DESIGN:
Intervention Model Description: Groups A, B and C are run sequentially.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part A, Group 1 (Active Comparator): Forearm stimulation during wake (study PART A) - electrode placement = volar surface of forearm, 2 electrodes (cathode and anode): Group 1 will receive forearm stimulation at 0.75 Hz with an oscillating direct current (DC) waveform while awake.
  Interventions: Device: transcranial electric stimulation
- Part A, Group 2 (Active Comparator): Forearm stimulation during wake (study PART A) - electrode placement = volar surface of forearm, 2 electrodes (cathode and anode): Group 2 will receive forearm stimulation at 0.75 Hz with a modified alternating current (AC) waveform while awake.
  Interventions: Device: transcranial electric stimulation
- Part A, Group 3 (Active Comparator): Forearm stimulation during wake (study PART A) - electrode placement = volar surface of forearm, 2 electrodes (cathode and anode): Group 3 will receive forearm stimulation at 3.0 Hz with an alternating current (AC) sinusoidal waveform while awake.
  Interventions: Device: transcranial electric stimulation
- Part B, Group 4 (Active Comparator): Scalp stimulation during sleep (study PART B) - bilateral electrode pairs placed on the upper forehead near the midline (F3 and F4) and adjacent to the ear in the mastoid region (M1 and M2). roup 4 will receive scalp stimulation at 0.75 Hz with an oscillating direct current (DC) waveform during sleep.
  Interventions: Device: transcranial electric stimulation
- Part B, Group 5 (Active Comparator): Scalp stimulation during sleep (study PART B) - bilateral electrode pairs placed on the upper forehead near the midline (F3 and F4) and adjacent to the ear in the mastoid region (M1 and M2). Group 5 will receive scalp stimulation at 0.75 Hz with a modified alternating current (AC) waveform during sleep.
  Interventions: Device: transcranial electric stimulation
- Part B, Group 6 (Active Comparator): Scalp stimulation during sleep (study PART B) - bilateral electrode pairs placed on the upper forehead near the midline (F3 and F4) and adjacent to the ear in the mastoid region (M1 and M2). Group 6 will receive scalp stimulation at 3.0 Hz with an alternating current (AC) sinusoidal waveform during sleep.
  Interventions: Device: transcranial electric stimulation
- Part C, Group 7 (Active Comparator): Pulsed Stimulation: Group 7 (Part C)will receive a series of brief stimulations of up to 500 millisecond duration and of up to 5 milliamperes of current, using either metal electrodes or sponge electrodes as stimulating electrodes.
  Interventions: Device: transcranial electric stimulation

INTERVENTIONS:
Device: transcranial electric stimulation — NeuroConn® DC Plus stimulator: the NeuroConn® stimulator can be programmed with specific frequencies of stimulation ranging from 0.5 to 500 Hz. This device is therefore appropriate for the present study to stimulate only at 0.75 or 3.0 Hz. Also, the NeuroConn only allows low current intensities to be chosen. The maximum current intensity that can be delivered with this stimulator is 5 milliamps.

SUMMARY:
Transcranial electrical stimulation (TES) utilizing weak electrical fields (<5 milliamps of current - as proposed in the present pilot study) is an extremely safe therapeutic technique in use for over 40 years. During that time, TES has never been associated with a serious adverse event in a research setting nor a serious reported adverse event in a clinical setting. The main side effect associated with TES is irritation of the skin beneath the electrodes (as is commonly found from similar preparations used for polysomnography). The purpose of this pilot study is to identify the type of electrode preparation that maximizes subject comfort during transdermal/transcranial electrical stimulation (TES) using the NeuroConn DC Plus Stimulator.

DETAILED DESCRIPTION:
In this study, volunteers will be divided into groups based on the nature of the stimulation waveform utilized (DC 0.75 Hz, modified AC 0.75 Hz, AC sinusoidal 3.0 Hz or pulsed stimulation of up to 500 ms duration). These waveforms were chosen based on the physiology of slow-wave sleep (SWS). Ultimately, the goal is to use TES during sleep to enhance the slow-wave activity (SWA) of sleep. Slow-wave sleep is characterized by two main frequency bands with differing underlying physiologies: (1) slow oscillation activity with a peak of 0.75 Hz, and (2) delta activity with a peak of approximately 3.0 Hz. Therefore, in future studies, the plan is to stimulate at one or both of these frequencies. The endogenous slow activity of the brain consists of electrical fields of "alternating current" with periods of relative cellular depolarization and periods of relative cellular hyperpolarization. The goal is to enhance this endogenous behavior with transcranial electrical stimulation at the two major slow- wave frequencies (0.75 Hz, 3.0 Hz), or using a pulsed stimulation paradigm to induce slow wave activity.

ELIGIBILITY:
Inclusion criteria - healthy adult men and non-pregnant, non-lactating women aged 18-39 years, inclusive.

Exclusion criteria - The following exclusion criteria apply to all volunteers, are consistent with those used in our other sleep studies, and are applied in this protocol in order to obtain a sample of volunteers who are likely to be representative of future study populations:

* Self-reported habitual nightly sleep amounts outside the target range of 6-9 hours (i.e., less than 6 hours per night or more than 9 hours per night, on average):
* Nighttime lights-out times earlier than 2100 hours on average during weeknights (Sunday through Thursday) for the past month
* Morning wake-up times later than 0900 on average during weekdays (Monday through Friday) for the past month.
* History of cardiovascular disease (to include but not limited to arrhythmias, valvular heart disease, congestive heart failure, history of sudden cardiac death or myocardial infarction)
* Reported habitual napping (> 3 times a week in conjunction with normal sleep habits)
* Resting blood pressure above 140/90
* Resting pulse > 110
* Neurologic disorder (to include but not limited to epilepsy or another seizure disorder, amnesia for any reason, hydrocephalus, MS, narcolepsy or other sleep disorders)
* Kidney disease
* History of psychiatric disorder requiring hospitalization or psychiatric medication for any length of time
* Beck Depression Inventory score of 14 or above
* Underlying pulmonary disease requiring daily inhaler use
* Regular nicotine use (or addiction) (defined as more than 1 cigarette or equivalent per week) within the last 1 year
* Positive nicotine/cotinine screen as determined by NicCheck™ I test strips
* Heavy alcohol use to be determined by the PI or his/her representative (minimum limit to define heavy alcohol use is 14 drinks per week)
* Use of other illicit drugs (to include but not limited to benzodiazepines, amphetamines, cocaine, marijuana)
* Known liver disease or liver abnormalities as determined by a laboratory test
* Self-reported history of caffeine use in excess of 400 mg (approximately 8 caffeinated sodas or 3-4 cups of coffee) per day on average
* Pregnancy (females)
* Inability to read and sign consent
* Use of certain medications (including use of vitamins or supplements), to be determined on a case-by-case basis by the examining study licensed physician.
* BMI ≥ 30 (Obese Class I or greater)
* The PI also maintains the prerogative to disqualify a volunteer if it is deemed that the volunteer's participation would be unsafe for the volunteer or staff or would be disruptive to study conduct.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2014-05-24 (Actual); Primary Completion 2029-02-12 (Estimated); Study Completion 2029-02-12 (Estimated)

PRIMARY OUTCOMES:
Sensation scale | Day 1
  participants indicate level of sensation on a scale from 1-10; Sensation Scale: 0 to 10 where 10 indicates experiencing severe discomfort; 0 indicates no discomfort
Erythema observation | Day 1
  observation of skin erythema following removal of electrodes: At baseline observation for presence of skin lesions/pathology; following stimulation observation of a change or no change in skin lesions/pathology from baseline

IPD SHARING:
Plan to Share IPD: No